CLINICAL TRIAL: NCT05583292
Title: The Effectiveness of ASA, SORT and Sarcopenia Indices in Estimating Mortality and Morbidity in Gastrointestinal Tumour Surgery
Brief Title: Mortality Predictions With Scorring Indices in Gastrointestinal Tumours
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Fethi Gultop, MD, Anesthesiology and Reanimation Specialist, Principal Investigator, Lecturer MD, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 01f
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Gastrointestinal Tumours
Keywords: ASA-PS; SORT; Sarcopenia; Mortality; Morbidity
MeSH Terms: conditions — Sarcopenia | interventions — 4-azidosalicylic acid-phosphatidylserine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ASA-PS — The American Society of Anesthesiologists classification of physical status (ASA PS) is a scale consisting of 6 classes showing the preoperative comorbidity of the patient.
Other: SORT — Surgical outcome risk tool (SORT) is a scale used to estimate patient preoperative mortality/ morbidity, measured from sortsurgery.com.
Other: Sarcopenia — Sarcopenia represents a loss of muscle strength and mass in older individuals and people who have tumors. Sarcopenia score is valuable in predicting preoperative mortality/ morbidity

SUMMARY:
The ASA-PS, SORT and Sarcopenia scores of the patients who will undergo surgery for a gastrointestinal tumor will be recorded. Thus, the correlation between preoperative indices and mortality/morbidity will be evaluated.

DETAILED DESCRIPTION:
ASA-PS values of patients who are planned to be operated due to gastrointestinal tumor will be recorded, then SORT (The Surgical Outcome Risk Tool) values will be calculated from sortsurgery.com. Sarcopenia measurements will be made by the radiologist from the abdomen CT at the L-3 level.

The pathology results of the patients will be recorded. Morbidity and mortality rates will be recorded in the short and long term.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* operation for gastrointestinal tumors

Exclusion Criteria:

* patient rejection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing gastrointestinal tumor surgery in a tertiary madical center
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2023-02-11 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
rate of mortality | 6 months after surgery
  death depending on the operation

CONTACTS AND LOCATIONS:
Overall Officials: fethi gültop, MD, Principal Investigator — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu City Hospital, Istanbul, Turkey (Türkiye)